CLINICAL TRIAL: NCT00895505
Title: Safety and Efficacy of a D-Dimer-Guided Strategy for Extension of Secondary Prophylaxis of Venous Thromboembolism - a Prospective and Randomized Management Trial
Brief Title: D-Dimer Guided Oral Anticoagulant Treatment (OAT)
Acronym: DDOAT2006
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Collaborators: German Research Foundation (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Prof. Dr. Bernd Pötzsch, Institut für Experimentelle Hämatologie und Transfusionsmedizin, Universitätsklinikum Bonn
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: DDOAT2006
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2009-05-08 (Estimated); Status verified 2009-05

CONDITIONS: Deep Venous Thrombosis
Keywords: DVT; Venous thromboembolism; D-Dimer; thrombophilia; secondary prophylaxis; secondary prophylaxis using oral anticoagulant treatment (OAT); higher risk of recurrence in patients showing increased levels; of D-Dimer after withdrawal of OAT; D-Dimer-based treatment
MeSH Terms: conditions — Venous Thrombosis; Venous Thromboembolism; Thrombophilia | interventions — Phenprocoumon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oral anticoagulants (Active Comparator): Experimental intervention: Extension of OAT in VTE patients showing high plasma levels of D-Dimer after end of routine secondary prophylaxis.
  Interventions: Drug: Phenprocoumon; Drug: Warfarin-Natrium
- 2 (No Intervention): Control: Withdrawal of OAT in VTE patients after end of routine secondary prophylaxis and receiving low molecular weight heparin in risk situations.

INTERVENTIONS:
Drug: Phenprocoumon — Phenprocoumon 3 mg, tablet, INR adjusted
  Arms: oral anticoagulants
Drug: Warfarin-Natrium — Warfarin-Natrium 5 mg, tablet, INR adjusted
  Arms: oral anticoagulants

SUMMARY:
This clinical trial will investigate the hypothesis that D-Dimer testing can be successfully used to tailor the duration of OAT in patients after an unprovoked episode of deep venous thrombosis (DVT) using a prospective, randomized, and controlled design.

DETAILED DESCRIPTION:
After a first episode of acute deep venous thrombosis (DVT) the risk of recurrence is relatively high and clinical consequences are important. Therefore, secondary prophylaxis using oral anticoagulant treatment (OAT) is usually established in these patients. This treatment very effectively reduces the risk of recurrences but induces an increased risk of bleeding. Major bleeding complications can be expected in ~2% patient-years. Therefore, current recommendations limit OAT to a period of 3 to 12 months. After stopping of OAT, however, ~10 % of patients with an initial episode of unprovoked DVT will develop a recurrent event within 1 year. This group of patients may benefit from prolonged OAT. The results of 2 independent observational studies showed a significantly higher risk of recurrence in patients showing increased levels of D-Dimer after withdrawal of OAT. D-Dimer is a biomarker that indicates fibrin formation followed by fibrinolysis. Based on these data we hypothesize that D-Dimer testing can be successfully used to tailor the duration of OAT in patients after an unprovoked episode of DVT. This clinical trial will investigate this hypothesis using a prospective, randomized, and controlled design.

ELIGIBILITY:
Inclusion Criteria:

To be enrolled in this study, patients must:

* have an objectively confirmed first episode of unprovoked VTE or of VTE during a minor transient risk factor. Minor transient risk factors include 6 weeks of estrogen therapy, prolonged air travel (i.e., > 6 hours), pregnancy, less marked leg injuries or immobilization without injury or surgical intervention
* be scheduled to receive oral anticoagulant treatment for at least 3 months
* be willing to be randomized
* be willing to participate for the full duration of the study

Exclusion Criteria:

* pregnancy or breast feeding
* contraindications against OAT (i.e., intracranial hemorrhage, subarachnoid hemorrhage, hemorrhagic stroke)
* age < 18 years
* presence of antiphospholipid antibodies or any other thrombophilic risk factor requiring long-term OAT (i.e., antithrombin deficiency, hereditary PC deficiency)
* poor patient compliance

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-02; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of objectively documented deep vein thrombosis (DVT) and/or pulmonary embolism (PE) | Duration of intervention per patient (24 months)

SECONDARY OUTCOMES:
Incidence and severity of signs and symptoms associated with OAT-induced bleeding measured using the World Health Organization (WHO) bleeding scale. | Duration of intervention per patient (24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Poetzsch, Professor, Principal Investigator — Institut für Experimentelle Hämatologie und Transfusionsmedizin, Universitätsklinikum Bonn
Locations (1):
- Institut für Experimentelle Hämatologie und Transfusionsmedizin, Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia, Germany